CLINICAL TRIAL: NCT01629914
Title: Executive Functioning and Mindfulness in Adults With ADHD Imaging
Brief Title: Executive Functioning and Mindfulness in Adults With Attention Deficit/Hyperactivity Disorder Imaging
Acronym: EFMImaging
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study close-out
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00037192
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Attention-deficit/Hyperactivity Disorder
Keywords: Attention-deficit/hyperactivity disorder; executive functioning; mindfulness meditation; magnetic resonance imaging; healthy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Mindfulness Meditation — 8-week, group-based mindfulness meditation intervention

SUMMARY:
The main purpose of this study is to evaluate changes in brain functioning using an MRI machine following mindfulness meditation training.

DETAILED DESCRIPTION:
The broad objective of this proposal is to identify functional neuroanatomical correlates of changes in executive brain functioning prior to and following an 8-week, group-based mindfulness meditation intervention within a group of 10 adults diagnosed with Attention-deficit/hyperactivity disorder (ADHD). Another group of 10 adults diagnosed with ADHD will be placed in the waitlist condition.

Our primary hypothesis is that adults with ADHD in the treatment group will exhibit improved performance on a series of executive functioning tasks and that exposure to task stimuli will correspond to changes in neural functioning following an 8-week, group-based mindfulness intervention. Brain responses will be measured using blood-oxygenation-level-dependent (BOLD) fMRI signal in brain regions associated with emotional and executive processes prior to and following treatment.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-50 years
* meet DSM-IV criteria for ADHD
* intellectual functioning ≥ 80 as assessed by an IQ screener
* generally healthy (i.e., no major medical problems)

Exclusion Criteria:

* major medical condition that would make participation unsafe (e.g., have pacemaker or other metallic implant), uncomfortable (e.g., chronic pain)
* claustrophobic, or abnormally afraid of closed-in places
* current drug use

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
change from baseline in blood-oxygenation-level-dependent (BOLD) fMRI signal | baseline and 8-weeks
  Participants will be scanned prior to and following an 8-week group-based mindfulness meditation intervention

CONTACTS AND LOCATIONS:
Overall Officials: John T Mitchell, Ph.D, Principal Investigator — Duke University